CLINICAL TRIAL: NCT01685736
Title: Ambulatory Versus Home Blood Pressure Monitoring in Obstructive Sleep Apnea
Acronym: OSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, George S. Stergiou, Associate Professor of Medicine and Hypertension, University of Athens
Other Study IDs: OSA
Record Dates: First submitted 2012-09-11; First posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Obstructive Sleep Apnoea; Hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Subjects referred to a sleep clinic had polysomnography (PSG), clinic BP measurements, 24-hour ABP monitoring and HBP monitoring using a device (Microlife WatchBP HomeN) that allows daytime (3 days, 2 duplicate readings/day) and automated nighttime BP measurement (3 nights, 3 readings/night).

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 65 years
* Suspected OSA
* Treated or untreated for hypertension

Exclusion Criteria:

* History of cardiovascular disease (heart failure, coronary heart disease, arrhythmia or stroke)
* History of asthma or chronic obstructive pulmonary disease (FEV1/FVC <70%)
* History of diabetes mellitus, collagen diseases and sarcoidosis
* Serum creatinine >1.6 mg/dl, proteinuria
* Previous treatment with CPAP
* Pregnancy or menstruation during the study
* Treatment with steroids, lithium or any other drugs affecting BP
* Change in antihypertensive treatment(if any) in the last 8 weeks before study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred to a sleep clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - First University Department of Respiratory Medicine, Sotiria Hospital, Athens
  - Hypertension Center, Third Department of Medicine, University of Athens, Greece, Athens